CLINICAL TRIAL: NCT01581580
Title: Deep Brain Stimulation Surgery for Movement Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110211; 11-N-0211
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-07-18

CONDITIONS: Parkinson's Disease; Essential Tremor; Dystonia
Keywords: Parkinson's Disease; Deep Brain Stimulation; Neurophysiology; Movement Disorder; Dystonia; Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia; Movement Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- treatment arm (Other): patients with Parkinson's Disease, dysonia, and essential tremor
  Interventions: Device: Medtronic Activa Tremor Control System; Procedure: Deep Brain Stimulation

INTERVENTIONS:
Device: Medtronic Activa Tremor Control System — Medtronic DBS Therapy delivers electrical stimulation to an area in the brain to help treat Parkinson's Disease, dystonia, and essential tremor.
Procedure: Deep Brain Stimulation — standard of care DBS surgery for patients with Parkinson's Disease, dystonia, and essential tremor

SUMMARY:
Background:

- Deep brain stimulation (DBS) is an approved surgery for certain movement disorders, like Parkinson's disease, that do not respond well to other treatments. DBS uses a battery-powered device called a neurostimulator (like a pacemaker) that is placed under the skin in the chest. It is used to stimulate the areas of the brain that affect movement. Stimulating these areas helps to block the nerve signals that cause abnormal movements. Researchers also want to record the brain function of people with movement disorders during the surgery.

Objectives:

* To study how DBS surgery affects Parkinson s disease, dystonia, and tremor.
* To obtain information on brain and nerve cell function during DBS surgery.

Eligibility:

- People at least 18 years of age who have movement disorders, like Parkinson's disease, essential tremor, and dystonia.

Design:

* Researchers will screen patients with physical and neurological exams to decide whether they can have the surgery. Patients will also have a medical history, blood tests, imaging studies, and other tests. Before the surgery, participants will practice movement and memory tests.
* During surgery, the stimulator will be placed to provide the right amount of stimulation for the brain. Patients will perform the movement and memory tests that they practiced earlier.
* After surgery, participants will recover in the hospital. They will have a followup visit within 4 weeks to turn on and adjust the stimulator. The stimulator has to be programmed and adjusted over weeks to months to find the best settings.
* Participants will return for followup visits at 1, 2, and 3 months after surgery. Researchers will test their movement, memory, and general quality of life. Each visit will last about 2 hours.

DETAILED DESCRIPTION:
Objective:

The objective of this protocol is to collect prospective physiology data related to DBS therapy and motor and cognitive function in people with medically refractory Parkinson's disease (PD), dystonia, and essential tremor (ET). All treatment under this protocol will be based on the current standard of care for DBS surgery.

Study Population:

Patients 18 years and older with medically refractory PD, dystonia and/or ET may participate in this study.

Study Design:

The treatment that is rendered in this protocol is standard of care for PD, dystonia, and ET. Patients confirmed to have medically refractory PD, dystonia or ET will be offered DBS. The therapeutic goal of this procedure is to implant chronically stimulating macroelectrodes in the basal ganglia or thalamic nuclei in order to alleviate the symptoms of PD, dystonia or ET. Pre- and post-operative imaging will be used to precisely localize electrode locations within the brain and will be correlated with measures of clinical efficacy and recorded intra-operative neural activity. Intra-operative microelectrode recordings, as well as micro- and macroelectrode electrical stimulation, will be used to confirm positioning of electrode leads. Intra-operative electrode recordings will also be used to investigate the neurophysiological mechanisms of deep brain stimulation and to explore the neural circuits underlying motor and cognitive processing in the basal ganglia. Intraoperative physiology will be used for clinical and research purposes. Patients will be followed for 3 months after the surgical procedure to determine effectiveness of DBS treatment.

Outcome Measures:

The primary goal of this protocol is to characterize motor and cognitive function in people receiving standard of care DBS surgery for movement disorders. Secondary measures include 1) radiographic correlation of DBS electrode position and clinical changes; and 2) neurophysiological mechanisms of DBS and motor and cognitive function in the basal ganglia.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, candidates must meet all the following criteria:

Be 18 years of age or older.

Able to provide informed consent.

Have a clinical diagnosis of one of the following as confirmed by the NIH movement disorders clinic team and the multi-disciplinary DBS surgical conference, and deemed as appropriate for the use of Deep Brain Stimulation therapy:

* idiopathic PD not adequately controlled with medication or
* primary dystonia that is medically refractory, or
* ET that is not adequately controlled by medications or constitutes a significant functional disability.

EXCLUSION CRITERIA:

Candidates will be excluded if they:

Are unable or unwilling to give informed consent to the research procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08-17 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
physiology and efficacy of DBS surgery for movement disorders | 3 months
  change in UPDRS III scale, Burke-Fahn-Marsden (BFM) scale, and Tremor Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Lau LM, Breteler MM. Epidemiology of Parkinson's disease. Lancet Neurol. 2006 Jun;5(6):525-35. doi: 10.1016/S1474-4422(06)70471-9. PMID 16713924
- [Background] DeLong MR. Primate models of movement disorders of basal ganglia origin. Trends Neurosci. 1990 Jul;13(7):281-5. doi: 10.1016/0166-2236(90)90110-v. PMID 1695404
- [Background] Alexander GE, Crutcher MD. Functional architecture of basal ganglia circuits: neural substrates of parallel processing. Trends Neurosci. 1990 Jul;13(7):266-71. doi: 10.1016/0166-2236(90)90107-l. PMID 1695401
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-N-0211.html